CLINICAL TRIAL: NCT06109259
Title: An Open-label, Randomized, 2x4 Crossover Study to Compare the Pharmacokinetics and Safety Following Administration of DWJ1567 and DWC202312 in Healthy Volunteers
Brief Title: Bioequivalence Study for the Safety and the Pharmacokinetics of DWJ1567 in Healthy Adult Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DWJ1567101
Record Dates: First submitted 2023-10-23; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DWJ1567 (Experimental): DWJ1567
  Interventions: Drug: DWJ1567
- DWC202312 (Active Comparator): DWC202312
  Interventions: Drug: DWC202312

INTERVENTIONS:
Drug: DWJ1567 — One tablet of DWJ1567
  Arms: DWJ1567
Drug: DWC202312 — One tablet of DWC202312
  Arms: DWC202312

SUMMARY:
This study aims to compare the pharmacokinetics and safety following administration of DWJ1567 and DWC202312 in healthy volunteers

DETAILED DESCRIPTION:
The study design is a Randomized, Open-label, Oral, Single-dose, Four-way crossover study. The patients were randomly assigned to each group. Primary endpoint was Cmax and AUCt of DWJ1567 and DWC202312. Secondary endpoints were AUCinf, Tmax, t1/2 of DWJ1567 and DWC202312.

ELIGIBILITY:
Inclusion Criteria:

* Over 19 year old

Exclusion Criteria:

* Galactose intolerance
* Lapp lactase deficiency

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-11-06 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Cmax,ss of DWJ1567 and DWC202312 | At pre-dose (0 hour), and post-dose 0 to 72 hour.
AUCt of DWJ1567 and DWC202312 | At pre-dose (0 hour), and post-dose 0 to 72 hour.

SECONDARY OUTCOMES:
AUCinf of DWJ1567 and DWC202312 | At pre-dose (0 hour), and post-dose 0 to 72 hour
Tmax of DWJ1567 and DWC202312 | At pre-dose (0 hour), and post-dose 0 to 72 hour
AUCt/AUCinf of DWJ1567 and DWC202312 | At pre-dose (0 hour), and post-dose 0 to 72 hour
t1/2 of DWJ1567 and DWC202312 | At pre-dose (0 hour), and post-dose 0 to 72 hour

CONTACTS AND LOCATIONS:
Locations (1):
- H Plus YANGJI Hospital, Seoul, South Korea